CLINICAL TRIAL: NCT01530789
Title: Evaluation of Paramedical Consultation in Type 1 Diabetic Patients in Telemedicine
Brief Title: Paramedical Consultation in Telemedicine
Status: Terminated | Type: Observational
Sponsor: Centre d'Etudes et de Recherche pour l'Intensification du Traitement du Diabète (Other)
Responsible Party: Sponsor
Other Study IDs: 2011-A00311-40
Record Dates: First submitted 2012-02-08; First posted 2012-02-10 (Estimated); Last update posted 2015-08-06 (Estimated); Status verified 2012-10

CONDITIONS: Type 1 Diabetic
Keywords: Telemedecine; Telemedecine nurse; Delegation of tasks; Type 1 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
Feasibility monocentrique opened study estimating the use of an electronic personalized educational plan (ePEP) for the follow-up by nurses of 50 patients diabetics type 1 during 6 months having an electronic pad.

ELIGIBILITY:
Inclusion Criteria:

* patient diabetic type 1
* patient with the electronic pad in a smartphone
* adults
* children between 12 and 17 years 11 months
* patient having signed the consent

Exclusion Criteria:

* patient diabetic type 2
* patient without the electronic pad in a smartphone
* children below 12 years old

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Diabetic type 1 patients with the electronic pad
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2011-05; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Percentage of patient using the system | 6 month
  The using of the system is estimated by the frequency of dose proposition by electronic pad

SECONDARY OUTCOMES:
satisfaction level of the patient and quality of life | 6 month
satisfaction level of physician | 6 month
  The satisfaction level of physician about the follow-up by e-PEP
satisfaction level of the telemedecin nurse | 6 month
  Evaluation of the satisfaction level of the telemedecin nurse about the follow-up by e-PEP